CLINICAL TRIAL: NCT00901563
Title: Gap Junction Potentiation of Endothelial Function With Rotigaptide in the Human Forearm Arterial Circulation - Effects of Ischaemia Induced Endothelial Dysfunction
Brief Title: Gap Junction Potentiation of Endothelial Function With Rotigaptide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: Chief Scientist Office of the Scottish Government (Other Government); NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: CZB/4/520/b
Record Dates: First submitted 2009-05-13; First posted 2009-05-14 (Estimated); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Vascular Disease; Heart Disease
Keywords: Gap Junctions; Rotigaptide; Ischaemia reperfusion; t-PA; Fibrinolysis; Endothelial function; Venous occlusion plethysmography
MeSH Terms: conditions — Vascular Diseases; Heart Diseases | interventions — rotigaptide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rotigaptide (Active Comparator): Prior to 20 mins of ischaemia induced by a blood pressure cuff inflated to 200 mmHg around the upper non-dominant arm, rotigaptide will be infused for 30mins. During the ischaemic period no drug will be infused but the infusion will be restarted once the blood pressure cuff has been deflated and blood flow returns to the limb.
  Interventions: Drug: Rotigaptide; Other: Forearm vascular study
- Saline (Placebo Comparator): Saline will be infused through-out the study.
  Interventions: Other: Forearm vascular study

INTERVENTIONS:
Drug: Rotigaptide — Prior to 20 mins of ischaemia induced by a blood pressure cuff inflated to 200 mmHg around the upper non-dominant arm, rotigaptide will be infused for 30mins. During the ischaemic period no drug will be infused but the infusion will be restarted once the blood pressure cuff has been deflated and blood flow returns to the limb.
  Arms: Rotigaptide
Other: Forearm vascular study — Forearm blood flow measured by venous occlusion plethysmography during interarterial infusion of substance P (2,4,8 pmol/min) or Acetylcholine (5, 10 , 20 micromol/min) . Venous blood sampling via cannula in antecubital fossa.

SUMMARY:
Hypothesis - Rotigaptide will improve endothelial function in the context of endothelial dysfunction.

The lining of blood vessels (endothelium) can react to hormones in the blood stream causing the blood vessel muscle to relax (vasodilatation) and allow more blood to flow. The nitric oxide and prostacyclin pathways are well documented in this process. However, evidence points to the existence of a third powerful relaxant called endothelium derived hyperpolarising factor (EDHF) but its identity and mechanism of action have proved elusive. As well as causing blood vessels to relax and more blood to flow, EDHF may be involved in the endothelium signaling, triggering release of a specialised clot dissolving factor called tissue plasminogen activator (t PA). t PA is important to ensure small clots, which are constantly being formed in the circulation, are rapidly dissolved and do not grow large enough to cause heart attacks and strokes.

Evidence points towards the requirement for 'gap junctions' in the mediation of EDHF responses. Gap junctions are specialised pores which allow small molecules and charge to pass between cells. They are found between endothelial cells and the underlying muscle of the blood vessel. A drug called Rotigaptide has been developed to cause gap junctions to open. It has been safely administered in healthy volunteers and is now in a Phase II drug trial. By opening gap junctions the investigators hypothesise that it could increase EDHF mediated activity and vasodilatation. It represents a useful tool with which to examine the role of gap junctions in EDHF activity in vivo.

Previously the investigators have demonstrated that rotigaptide does not contribute to endothelial function in healthy volunteers. The investigators now wish to examine the effect of rotigaptide in conditions of endothelial dysfunction. By limiting the blood flow to the arm for 20mins the ability of the blood vessel to vasodilate is impaired. By administering an intra-arterial rotigaptide infusion the investigators want to assess any functional preservation.

DETAILED DESCRIPTION:
BACKGROUND The endothelium plays a pivotal role in the control of vascular tone and is responsible for the local release of profibrinolytic factors. Nitric oxide (NO), the original endothelium-derived relaxing factor, and prostacyclin (PGI2) have now been well characterised. The elucidation of their roles in vascular physiology and pathophysiology has been fundamental to recent advances in the treatment and prevention of many cardiovascular diseases. Whilst these factors are of major importance, evidence points to the existence of a third powerful vasodilator called endothelium-derived hyperpolarising factor (EDHF).

Endothelium-dependent vasodilatation -

After blockade of both NO and PGI2, a substantial degree of endothelium-dependent vasodilatation is still observed and is attributed to EDHF. Despite almost two decades of research and debate, the exact nature of EDHF and its mechanism of action remain unclear. Consistently, EDHF's role as a vasodilator is most prominent in the smaller resistance arteries that are responsible for the control of systemic blood pressure and local organ perfusion. As well as its involvement in physiological processes, alterations in EDHF activity may contribute to the vascular effects of the myriad of conditions either caused by, or resulting in, endothelial dysfunction. However, the lack of understanding of EDHF has precluded its direct manipulation as a specific therapeutic target.

Endogenous fibrinolysis -

In addition to its function in the control of vascular tone, there is evidence to suggest that EDHF may be responsible for the endothelial release of the pro-fibrinolytic factor, tissue-type plasminogen activator (t-PA).

Thrombus formation and dissolution is a continuous process in the vasculature and is regulated by dynamic interactions between pro-coagulant and pro-fibrinolytic factors. Endogenous fibrinolysis is determined by the relative balance between the acute local release of t-PA from the endothelium and its subsequent inhibition by plasma plasminogen activator inhibitor type 1 (PAI-1). In the presence of an imbalance in the fibrinolytic system, subclinical microthrombi on the surface of atherosclerotic plaques may propagate and ultimately lead to arterial occlusion and tissue infarction.

The mechanisms via which t-PA release is mediated are incompletely understood. Bradykinin, an endogenous endothelium-dependent vasodilator, causes the endothelial release of t-PA. However, Brown et al have demonstrated that inhibition of prostacyclin and nitric oxide synthesis does not diminish bradykinin mediated endothelial t-PA release in the human forearm. Therefore, they suggest that EDHF is responsible for the endothelial release of t-PA but, to date, this hypothesis has not been adequately addressed.

Gap Junctions -

Gap junctions are found at points of cell-cell contact where they form an aqueous pore through which small hydrophilic molecules and ionic charge may pass. Each gap junction comprises two hemichannels, or connexons that are composed of six connexin (Cx) subunits. Although each connexon may be composed of a mix of connexin subtypes, Cx37, Cx40 and Cx43 are particularly associated with mammalian endothelium and vascular smooth muscle.

The case for a pivotal role of gap junctions in the EDHF phenomenon has strengthened. Gap junction plaques are most abundant in small resistance arteries and their distribution is proportional to the magnitude of the EDHF-mediated response. These topographical data have been extrapolated to argue for a direct link between gap junctions and EDHF. Furthermore, murine knockout models provide direct evidence for a role of gap junctions and specific connexins in the control of vascular tone.

Potentiation of Communication via Gap Junctions -

Rotigaptide (ZP-123) is a novel hexapeptide (Ac-D-Tyr-D-Pro-D-Hyp-Gly-D-Ala-Gly-NH2), originally developed as an antiarrythmic agent it has now been safely administered to healthy humans as a six day continuous infusion of up to 20 mg (0.30 mmol) per day and is now in Phase II clinical trials. It has been shown to promote electrical coupling between ventricular myocytes by increasing gap junction conductance potentially via alterations in the phosphorylation status of Cx43 and it increases the number of gap junctions in the ischaemic myocardium It potentiates gap junction-mediated dye transfer via Cx43 expressing HeLa cells but not via Cx26 or Cx32 but its effects on electrical conduction and dye transfer via Cx37 and Cx40, the other major vascular connexins, have yet to be assessed. However, we have recently shown that Cx43 is required for the mediation of EDHF vasodilatation of human subcutaneous resistance vessels.

We have recently demonstrated that rotigaptide does not enhance endothelium-dependent or independent forearm arterial vasodilatation in healthy volunteers. However there may be a role for potentiating gap junctions under some circumstances. In animal models of myocardial infarction those treated with rotigaptide had significantly reduced infarction sizes. Endothelial dysfunction is central to the pathophysiology of diabetes and is responsible for the vascular complications associated with this condition. In animal models of diabetes reduced expression of connexins has been demonstrated with blunted response to EDHF, suggesting a link between endothelial dysfunction and gap junctions.

Endothelial dysfunction can be mimicked in vivo with brief periods of ischaemia, resulting in a reduced response to endothelium-dependant vasodilators. In the forearm arterial circulation, we will test the hypothesis that rotigaptide-induced enhancement of communication via gap junctions attenuates ischaemic endothelial dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers aged between 18-64 years.

Exclusion Criteria:

* Lack of informed consent
* Age <18 or >64 years
* Current involvement in a clinical trial
* Clinically significant comorbidity: heart failure, hypertension, known hyperlipidaemia, diabetes mellitus, asthma, coagulopathy or bleeding disorders*
* Smoker*
* Current intake of aspirin, other non steroid anti inflammatory medications or vasodilators*
* Recent infective/inflammatory condition*
* Women of child bearing age
* Recent blood donation (preceding three months) *All cause confounding effects on vascular/endothelial function.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2009-03 (Actual); Primary Completion 2015-08-03 (Actual); Study Completion 2015-08-03 (Actual)

PRIMARY OUTCOMES:
Change in Substance P and ACh vasodilatation caused by potentiation of gap junction communication with Rotigaptide in the context of endothelial dysfunction | Vasodilatation will be assesed before and after ischaemic periods

SECONDARY OUTCOMES:
Change in Substance P induced t PA release caused by potentiation of gap junction communication with Rotigaptide in the context of endothelial dysfunction | Venous blood samles will be taken at regular time points throught the protocol

CONTACTS AND LOCATIONS:
Overall Officials: David E Newby, MD, Study Director — University of Edinburgh
Locations (1):
- Clincial Research Facility, Royal Infirmary of Edinburgh, 51 Little France Cresc, Edinburgh, United Kingdom

REFERENCES:
- [Result] Pedersen CM, Venkatasubramanian S, Vase H, Hyldebrandt JA, Contractor H, Schmidt MR, Botker HE, Cruden NL, Newby DE, Kharbanda RK, Lang NN. Rotigaptide protects the myocardium and arterial vasculature from ischaemia reperfusion injury. Br J Clin Pharmacol. 2016 Jun;81(6):1037-45. doi: 10.1111/bcp.12882. Epub 2016 Mar 10. PMID 26750458